CLINICAL TRIAL: NCT02201173
Title: Health Outcomes After Locomotor Training in Spinal Cord Injury Across the NeuroRecovery Network
Brief Title: Health Outcomes After Locomotor Training in Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Ohio State University (Other); Kessler Institute for Rehabilitation (Industry); TIRR Memorial Hermann (Other); University of Louisville (Other); Craig Hospital (Other)
Responsible Party: Principal Investigator, Sue Ann Sisto, Professor of Health Sciences and Research Director, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 376696
Record Dates: First submitted 2014-07-02; First posted 2014-07-25 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injuries; Spinal Cord Trauma
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Locomotor Training (Experimental)
  Interventions: Behavioral: Locomotor Training

INTERVENTIONS:
Behavioral: Locomotor Training — Progressive retraining in functional skills including balance, transfers, activities of daily living and ambulation. Compliance to eliminate or minimize lower limb orthotics is also expected to optimize sensory input to the spinal cord and promote optimal recovery. Intensive therapy occurs in all three environments 5 times/ week for 90 minutes

SUMMARY:
People with spinal cord injury (SCI) suffer from secondary health conditions that can result in undue physical challenges and impact participation in activities in everyday life. Locomotor Training (LT) has been shown to demonstrate improvements in balance and walking function in both the animal and humans by reactivating spinal circuits through intensive therapy of muscles below the level of the injury. However, it is not known if LT also has beneficial health effects and it is the focus of this study proposed to be undertaken at Stony Brook University (SBU) as the lead site. LT is thought to produce activation of spinal networks to help recover balance and walking after SCI and may correspond with improvements in health measures such as bladder function, breathing capacity, cholesterol and other cardiac risk factors markers, and the ability to stand upright without drops in blood pressure resulting in a sensation of dizziness. LT takes place on a treadmill with the body weight supported in a harness, while walking overground and with the practice of key exercises in the home and community. The emphasis is on loading the body through the legs without braces and other devices except where necessary to function at home. The overall objective of this study to capture and analyze health outcome data collected on 80 patients enrolled in the 7 NeuroRecovery Network (NRN) clinics in the USA who receive LT. The NRN is funded by the Christopher and Dana Reeve Foundation and the CDC to implement LT for people with SCI. The purpose of this application is to leverage the NRN funding, that provides support for LT and standardized outcome measures, to generate further knowledge on health outcomes after LT for individuals with SCI. The proposed project will be accomplished through the utilization of staff at each of the 6 NRN sites, lead by the study principal investigator and the lead clinical research coordinator at SBU. They will ensure the data are captured before and after LT in a standardized manner, at the correct time and entered into a de-identified database. The study hypotheses are that after LT, compared to before, patients with SCI will improve lipid profiles and insulin factors as measured by fasting blood tests; respiratory function as measured by specialized but easy to use breathing equipment; and blood pressure and heart rate during a maneuver to test for responses to abrupt changes in posture. The relevance of this proposal is that it will help to determine if there is an association between an intensive activity- based intervention (LT) and improvements in health and will be used to form the basis for a larger randomized clinical trial and clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are classified as AIS C and D must have some lower limb movement or visible voluntary contraction and the capacity to generate a lower limb reciprocal alternating flexion/extension stepping pattern in the step training environment using body weight support on a treadmill with manual facilitation.
* Patients with AIS A and B need to be able to stand in the BWS harness system without orthostatic hypotension for at least 1 minute.

Exclusion Criteria:

* Anti-spasticity medication except night time dose.
* The use of chemodenervation for spasticity will be avoided for the 3 months prior to NRN admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Blood Assays | Baseline and after 80 sessions of Locomotor Training (LT). If continuous sessions are attended then 5d X 16 weeks or 4 months = 80 sessions.
  Study supplements the Locomotor Training program sponsored by the NeuroRecovery Network except for this new study where blood is drawn before and after Locomotor Training (LT)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Craig Hospital, Englewood, Colorado
  - Frazier Rehab, Louisville, Kentucky
  - Rehabilitation Research and Movement Performance Lab, Stony Brook, New York